CLINICAL TRIAL: NCT06759545
Title: Effect of Extra Virgin Olive Oil Addition in the Diet of Women with Higher Risk for Preeclampsia - Interventional Pilot Study
Brief Title: An Interventional Pilot Study on the Effect of Extra Virgin Olive Oil on Women with Preeclampsia Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yaniv Ovadia (Other)
Responsible Party: Sponsor-Investigator, Yaniv Ovadia, Dr Yaniv S. Ovadia RD PhD, Barzilai Medical Center
Organization: Barzilai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0049-24-BRZ
Record Dates: First submitted 2024-12-17; First posted 2025-01-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Preeclampsia (PE) Risk
Keywords: Extra virgin olive oil from early harvested olives; preeclampsia; FMS-like tyrosine kinase 1; plasma hydroxytyrosol; dietary intervention; point Mediterranean Diet Adherence Screener; prevention
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EVOOEH arm (Experimental): Daily addition of 42 ml (three tablespoon) at each morning of EVOOEH to MOH recommendations for 4 weeks (n=78).
  Interventions: Other: Dietary MOH recommendations and daily addition of 42 ml (three tablespoon) at each morning of EVOOEH
- Control arm (Other): MOH recommendations for 4 weeks (n=78).
  Interventions: Other: Dietary MOH recommendations

INTERVENTIONS:
Other: Dietary MOH recommendations and daily addition of 42 ml (three tablespoon) at each morning of EVOOEH — Dietary intervention study: high-risk pregnant women receiving a link to MOH general dietary recommendations for pregnancy (MOH recommendations) with addition of three tablespoon (42 ml) EVOOEH (up to 0.8% free acidity) per day at each morning for four weeks during the first half of pregnancy (gestational ages between 8 to 16 weeks)
  Arms: EVOOEH arm
Other: Dietary MOH recommendations — Dietary intervention study: high-risk pregnant women receiving a link to MOH general dietary recommendations for pregnancy (MOH recommendations) for four weeks during the first half of pregnancy (gestational ages between 8 to 16 weeks)
  Arms: Control arm

SUMMARY:
This study explores the potential benefits of Extra Virgin Olive Oil from early harvested olives (EVOOEH) in reducing the risk of preeclampsia (PE) in high-risk pregnant women. EVOO, particularly EVOOEH, is rich in antioxidant compounds, including polyphenols, which may help improve vascular health and reduce oxidative stress, potentially preventing complications like PE. The hypothesis is that EVOOEH may reduce microvascular damage, improve placentation, and prevent dysglycemia, ultimately lowering the risk of PE and gestational diabetes mellitus (GDM).

The primary objective of this intervention is to evaluate the effect of EVOOEH on PE incidence during pregnancy, specifically assessing the impact on markers of PE, GDM, and other pregnancy-related outcomes. The study is designed as an interventional, randomized, parallel-assignment dietary trial involving 156 pregnant women at high risk for PE, aged 18 to 45. Participants will receive either a daily dose of 42 ml (three tablespoons) of EVOOEH or the Ministry of Health (MOH) general dietary recommendations for pregnancy for four weeks, starting between 8 to 16 weeks of gestation.

The study arms are as follows:

EVOOEH arm: Participants will consume 42 ml of EVOOEH daily along with MOH dietary recommendations for four weeks (n=78).

Control arm: Participants will follow only the MOH dietary recommendations for four weeks (n=78).

The intervention will occur alongside low-dose aspirin prophylaxis for PE prevention, as recommended by guidelines for women at high risk. Key compliance markers include adherence to a Mediterranean diet as measured by the Mediterranean Diet Adherence Screener (MEDASIS) and hydroxytyrosol levels in maternal blood. The study will mask data analysis to minimize bias.

The primary outcome measures are maternal glucose challenge test (GCT) results and the serum soluble FMS-like tyrosine kinase 1/placental growth factor (sFlt-1/PlGF) ratio at the end of the intervention. Secondary outcomes include the incidence of GDM, PE, cesarean sections, preterm delivery, small for gestational age (SGA) births, blood pressure measurements, gestational age at delivery, and any relevant data available from participants' medical records.

Eligibility criteria include pregnant women with risk factors for PE such as a history of PE, chronic hypertension, obesity, or diabetes, among others, and a gestational age between 8 to 16 weeks. Exclusion criteria involve low-risk pregnancies or women who refuse participation.

Blood samples will be collected to assess 25-hydroxyvitamin D (25(OH)D), hydroxytyrosol (HT), and the sFlt-1/PlGF ratio. Laboratory analyses will be conducted at Barzilai University Medical Center and the Weizmann Institute of Science. This study seeks to determine whether EVOOEH's higher polyphenol content compared to standard EVOO can offer additional protective benefits against PE and related complications in high-risk pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with clinical risk factors for PE [previous PE, primigravida, chronic hypertension, chronic renal disease, autoimmune disease (systemic lupus erythematosus, antiphospholipid antibody syndrome), overweight (BMI>30), obesity (BMI>35), morbid obesity (BMI>40), presentational diabetes (type 1 or type 2), multiple pregnancy].
* gestational ages of 8 to 16 weeks attending Barzilai University Medical Center at Ashkelon (BUMCA).

Exclusion Criteria:

• Refusing enrollment or participation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2027-01-07 (Estimated); Study Completion 2028-01-07 (Estimated)

PRIMARY OUTCOMES:
sFlt-1/PlGF ratio | 4 weeks
  Post intervention serum sFlt-1/PlGF ratio at the end of intervention.
GCT result | 4 weeks
  Post intervention maternal GCT result at the end of intervention.

SECONDARY OUTCOMES:
SBP | At recruitment and approximately 4 weeks post intervention initiation
  Maternal systolic diastolic blood pressure
DBP | At recruitment and approximately 4 weeks post intervention initiation
  Maternal diastolic diastolic blood pressure
PE | From intervention to delivery
  PE diagnosis
GDM | From intervention to delivery
  GDM diagnosis
CS | At delivery
  Cesarean section incidence
Preterm | At birth
  Preterm incidence
SGA | At birth
  SGA incidence
Birthweight percentile | At birth
  Newborn adjusted with percentile

CONTACTS AND LOCATIONS:
Overall Officials: Dr Yaniv S. Ovadia, RD PhD, Study Director — Barzilai University Medical Center Ashkelon
Locations (1):
- Barzilai University Medical Center, Ashkelon, Ashkelon District, Israel

IPD SHARING:
Plan to Share IPD: No